CLINICAL TRIAL: NCT03888365
Title: An Observational Study to Characterize Patient Global Impression Questions for Activity-induced Symptoms in Patients With Pulmonary Arterial Hypertension (PAH)
Brief Title: Patient Global Impression Questions for Activity-Induced Symptoms in Participants With PAH
Acronym: PRN
Status: Completed | Type: Observational
Sponsor: United Therapeutics (Industry)
Collaborators: Lung Biotechnology PBC (Industry)
Responsible Party: Sponsor
Other Study IDs: RIN-PRN-201
Record Dates: First submitted 2019-03-18; First posted 2019-03-25 (Actual); Results first posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-02

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Hypertension; Treprostinil; Pulmonary Hypertension; Lung Diseases
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension; Hypertension, Pulmonary; Lung Diseases | interventions — treprostinil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort A: Treprostinil: Participants who are currently prescribed and using inhaled treprostinil for the treatment of PAH.
  Interventions: Drug: Treprostinil
- Cohort B: Non-Treprostinil PAH Medications: Participants who are taking other PAH medications (instead of inhaled treprostinil).
  Interventions: Drug: Non-Treprostinil PAH Medications

INTERVENTIONS:
Drug: Treprostinil — Treprostinil treatment will be at the discretion of the participant's physician, and determined on an individual basis.
  Groups: Cohort A: Treprostinil
Drug: Non-Treprostinil PAH Medications — Non-treprostinil treatment will be at the discretion of the participant's physician, and determined on an individual basis.
  Groups: Cohort B: Non-Treprostinil PAH Medications

SUMMARY:
This is an observational, multicenter, single-day, Phase 2 study. This study will include a 14-day Screening Period and Study Day 1 clinic visit. Participants will be required to perform an activity to induce symptoms of PAH, and participants' severity of self-reported symptoms of PAH will be measured from pre-activity, immediately after the activity, and through the 30-minute recovery. Participants will be asked about their PAH symptoms using 3 PGI-S questions that address their overall PAH symptoms, shortness of breath, and physical fatigue.

DETAILED DESCRIPTION:
This is an observational, multicenter, single-day, Phase 2 study. This study will include a 14-day Screening Period and Study Day 1 clinic visit. Participants will be required to perform an activity to induce symptoms of PAH, and participants' severity of self-reported symptoms of PAH will be measured from pre-activity, immediately after the activity, and through the 30-minute recovery. Participants will be asked about their PAH symptoms using 3 Patient Global Impression of Severity (PGI-S) questions that address their overall PAH symptoms, shortness of breath, and physical fatigue.

PAH symptoms will be induced via the Incremental Shuttle Walk Test (ISWT). The ISWT used in this study required the participant to walk back and forth on a 10-meter course. The total number of shuttles completed by a participant during the Screening ISWT will be the maximum targeted for that participant during the remaining ISWTs in the study.

After Screening, participants will be assigned to 1 of 2 cohorts based on PAH medications as prescribed by their physician: Cohort A will include participants who are currently prescribed and using inhaled treprostinil for the treatment of PAH and Cohort B will include participants who are taking other PAH medications (instead of inhaled treprostinil).

The study also includes 2 periods. One period for participants in Cohort A (Treprostinil Users), included an ISWT initiated within 30 minutes of the previous dose (expected peak level) and the other period included an ISWT within 3 to 4 hours of the previous dose of inhaled treprostinil (expected trough level). Participants in Cohort B (Non-Treprostinil Users), an ISWT will be initiated approximately 4 hours after the morning dose of PAH medication (Period 1) and an ISWT initiated at least 1 hour following completion of the previous ISWT (Period 2). Participants will be provided at least a 1-hour period for rest between ISWTs (until participant feels they are rested enough to perform again at their baseline level) prior to Period 2 assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Participant voluntarily gives informed consent to participate in the study.
2. Males and females aged 18 years and above at the time of informed consent.
3. Established primary diagnosis of PAH that is either idiopathic or familial PAH (WHO Group 1), collagen vascular disease associated PAH, PAH associated with HIV infection, PAH induced by anorexigens/toxins, or PAH associated with repaired congenital systemic-to-pulmonary shunts (repaired ≥1 years).
4. Participant is deemed WHO Functional Class 1, 2, or 3.
5. Participant has shortness of breath upon exertion (exhibits a ≥1-point change in Borg dyspnea score) as assessed by the ISWT and a minimum completion of 3 shuttles (30 meters) of the ISWT. Participant may have other symptoms as well.
6. Participant is on stable dose of all FDA-approved PAH treatments (exceptions are anticoagulants and diuretics) for at least 60 days prior to Screening.
7. In the opinion of the Investigator, the participant can communicate effectively with study personnel, and is considered reliable, willing, and likely to be cooperative with protocol requirements.

Exclusion Criteria:

1. The participant is known to be pregnant or nursing.
2. The participant has PAH related to any condition not covered under inclusion criteria, including, but not limited to, pulmonary venous hypertension, pulmonary venoocclusive disease, pulmonary capillary hemangiomatosis, chronic thromboembolic pulmonary hypertension, or other conditions under WHO Group 2, 3, 4, and 5 classifications.
3. The participant has evidence of clinically significant left-sided heart disease (including, but not limited to, left ventricular ejection fraction <40%, left ventricular hypertrophy) or clinically significant cardiologic conditions, such as congestive heart failure, coronary artery disease, or valvular heart disease.
4. The participant has any form of congenital heart disease (repaired or unrepaired; other than a patent foramen ovale).
5. The participant has any ambulatory or orthopedic limitations that would interfere with the ability to perform the activity.
6. The participant has been hospitalized within 30 days of Screening.
7. Current use of prostacyclin analogs/agonists, except inhaled treprostinil, for the treatment of PAH.
8. Use of any other investigational drug/device, or participation in any investigational study with therapeutic intent within 30 days of Screening (concurrent participation in registry studies is allowed).
9. Any other clinically significant illness that, in the opinion of the Investigator, might put the participant at risk of harm during the study or might adversely affect the interpretation of the study data.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Males and females aged 18 years and above with a diagnosis of PAH that is either idiopathic or familial PAH (World Health Organization [WHO] Group 1), collagen vascular disease associated PAH, PAH associated with human immunodeficiency virus (HIV) infection, PAH induced by anorexigens/toxins, or PAH associated with repaired congenital systemic-to-pulmonary shunts (repaired ≥1 years).
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-09-19 (Actual); Study Completion 2019-09-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Cedars-Sinai Medical Center, Beverly Hills, California
  - Santa Barbara Pulmonary Associates, Santa Barbara, California
  - St. Francis Sleep, Allergy & Lung Institute, Clearwater, Florida
  - Pulmonary & Critical Care of Atlanta, Atlanta, Georgia
  - Kentuckiana Pulmonary Associates, Louisville, Kentucky
  - Pulmonary Health Physicians, PC, Fayetteville, New York
  - The Mount Sinai Hospital, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Rhode Island Hospital, Providence, Rhode Island

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study included a 14-day Screening Period and Day 1 clinic visit. Participants performed a Incremental Shuttle Walk Test (ISWT) to induce symptoms of Pulmonary Arterial Hypertension (PAH). The ISWT required participants to walk back and forth on a 10-meter course. Total number of shuttles completed by a participant during the Screening ISWT was the maximum targeted for the participant for remaining study ISWTs. Study also included 2 periods/cohort. There was ≥1-h rest period between ISWTs.
Pre-assignment Details: The 2 periods for Cohort A: an ISWT initiated at 30 minutes (m) of previous dose (the expected peak level period) and an ISWT initiated at 3-4 hours (h) of previous dose of inhaled treprostinil (the expected trough level period). The 2 periods for Cohort B: an ISWT initiated at ~4h after morning dose of PAH medication (Period 1) and an ISWT initiated at ≥1h following completion of previous ISWT (Period 2). Peak and trough levels are the highest and lowest concentrations of a drug in plasma.
Groups:
- Cohort A: Treprostinil: Participants who were currently prescribed and using inhaled treprostinil for the treatment of PAH.
- Cohort B: Non-Treprostinil PAH Medications: Participants who were taking other PAH medications (instead of inhaled treprostinil).
Period: Cohort A Peak Level/Cohort B Period 1
Arm/Group | Cohort A: Treprostinil | Cohort B: Non-Treprostinil PAH Medications
Started (All Participants: Participants who consented to the study protocol.) | 20 | 23
Safety Population (All participants who initiated an ISWT at Screening.) | 20 | 23
Completed | 20 | 23
Not Completed | 0 | 0
Period: Rest - At Least 1 h
Arm/Group | Cohort A: Treprostinil | Cohort B: Non-Treprostinil PAH Medications
Started | 20 | 23
Completed | 20 | 23
Not Completed | 0 | 0
Period: Cohort A Trough Level/Cohort B Period 2
Arm/Group | Cohort A: Treprostinil | Cohort B: Non-Treprostinil PAH Medications
Started | 20 | 23
Completed | 20 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All Participants: Participants who consented to the study protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Treprostinil | Cohort B: Non-Treprostinil PAH Medications | Total
Number analyzed (Participants) | 20 | 23 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (8.69) | 55.9 (13.14) | 58.3 (11.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 33
  Male | 4 | 6 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 19 | 21 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 14 | 18 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Patient Global Impression of Severity (PGI-S) Score in Cohort A Participants at Approximately 30 Minutes of Previous Dose of Inhaled Treprostinil (the Expected Peak Level) on Day 1
Description: A global index that consists of 3 questions to which participants will rate the severity of 1) their PAH symptoms, 2) shortness of breath (SOB), and 3) fatigue. The minimum and maximum range of scores for each of the 3 individual questions was 1-5, with severity scale choices of 1=Not present, 2=Mild, 3=Moderate, 4=Severe, and 5=Very Severe. A higher score indicated worse outcome. The Baseline is defined as the average respective severity rating measured at 15 minutes and 0 minute prior to the ISWT. In the case of a single, missing severity rating measured pre-ISWT, the other non-missing single severity rating would be used as baseline value. Only participants with both a measurement at baseline and at the given post-baseline visit are summarized. Change from Baseline = Post-Baseline value - Baseline value. Peak levels are the highest concentrations of a drug in plasma.
Time Frame: Baseline, Approximately 30 m of previous dose of inhaled treprostinil (the expected peak level) on Day 1
Population: All Participants: Participants who consented to the study protocol. Data for participants in Cohort A who included an ISWT initiated at 30 m of previous dose (expected peak level) are presented.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Cohort A: Treprostinil
Number analyzed (Participants) | 20
scores on a scale
  PAH, Baseline | 1.25 (0.47)
  PAH, Change at 30 m of previous dose of inhaled treprostinil (expected peak level) on Day 1 | 1.65 (0.80)
  SOB, Baseline | 1.15 (0.33)
  SOB, Change at 30 m of previous dose of inhaled treprostinil (expected peak level) on Day 1 | 1.90 (0.80)
  Fatigue, Baseline | 1.30 (0.55)
  Fatigue, Change at 30 m of previous dose of inhaled treprostinil (expected peak level) on Day 1 | 1.40 (0.95)

2. Primary Outcome: Change From Baseline in PGI-S Score in Cohort A Participants at Approximately 3-4 Hours of Previous Dose of Inhaled Treprostinil (the Expected Trough Level) on Day 1
Description: A global index that consists of 3 questions to which participants will rate the severity of 1) their PAH symptoms, 2) SOB, and 3) fatigue. The minimum and maximum range of scores for each of the 3 individual questions was 1-5, with severity scale choices of 1=Not present, 2=Mild, 3=Moderate, 4=Severe, and 5=Very Severe. A higher score indicated worse outcome. The Baseline is defined as the average respective severity rating measured at 15 minutes and 0 minute prior to the ISWT. In the case of a single, missing severity rating measured pre-ISWT, the other non-missing single severity rating would be used as baseline value. Only participants with both a measurement at baseline and at the given post-baseline visit are summarized. Change from Baseline = Post-Baseline value - Baseline value. Trough levels are the lowest concentrations of a drug in plasma.
Time Frame: Baseline, Approximately 3-4 h of previous dose of inhaled treprostinil (the expected trough level) on Day 1
Population: All Participants: Participants who consented to the study protocol. Data for participants in Cohort A who included an ISWT initiated at 3-4 h of previous dose of inhaled treprostinil (expected trough level) are presented.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Cohort A: Treprostinil
Number analyzed (Participants) | 20
scores on a scale
  PAH, Baseline | 1.10 (0.31)
  PAH, Change at 3-4 h of previous dose of inhaled treprostinil (expected trough level) on Day 1 | 1.75 (0.79)
  SOB, Baseline | 1.10 (0.31)
  SOB, Change at 3-4 h of previous dose of inhaled treprostinil (expected trough level) on Day 1 | 1.85 (0.93)
  Fatigue, Baseline | 1.25 (0.44)
  Fatigue, Change at 3-4 h of previous dose of inhaled treprostinil (expected trough level) on Day 1 | 1.50 (1.15)

3. Primary Outcome: Change From Baseline in PGI-S Score in Cohort B Participants at Approximately 4 Hours After Morning Dose of Non-Treprostinil PAH Medication (Period 1) on Day 1
Description: A global index that consists of 3 questions to which participants will rate the severity of 1) their PAH symptoms, 2) SOB, and 3) fatigue. The minimum and maximum range of scores for each of the 3 individual questions was 1-5, with severity scale choices of 1=Not present, 2=Mild, 3=Moderate, 4=Severe, and 5=Very Severe. A higher score indicated worse outcome. The Baseline is defined as the average respective severity rating measured at 15 minutes and 0 minute prior to the ISWT. In the case of a single, missing severity rating measured pre-ISWT, the other non-missing single severity rating would be used as baseline value. Only participants with both a measurement at baseline and at the given post-baseline visit are summarized. Change from Baseline = Post-Baseline value - Baseline value.
Time Frame: Baseline, Approximately 4 h after morning dose of non-treprostinil PAH medication (Period 1) on Day 1
Population: All Participants: Participants who consented to the study protocol. Data for participants in Cohort B who included an ISWT initiated at 4 h after morning dose of non-treprostinil PAH medication (Period 1) on Day 1 are presented.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Cohort B: Non-Treprostinil PAH Medications
Number analyzed (Participants) | 23
scores on a scale
  PAH, Baseline | 1.22 (0.39)
  PAH, Change at 4 h after morning dose of non-treprostinil PAH medication (Period 1) on Day 1 | 1.74 (0.90)
  SOB, Baseline | 1.17 (0.36)
  SOB, Change at 4 h after morning dose of non-treprostinil PAH medication (Period 1) on Day 1 | 1.78 (0.78)
  Fatigue, Baseline | 1.17 (0.36)
  Fatigue, Change at 4 h after morning dose of non-treprostinil PAH medication (Period 1) on Day 1 | 1.61 (1.07)

4. Primary Outcome: Change From Baseline in PGI-S Scores in Cohort B Participants With an ISWT at Least 1 h Following Completion of Previous ISWT (Period 2) on Day 1
Description: as for outcome 3
Time Frame: Baseline, At least 1 h following completion of previous ISWT (Period 2) on Day 1
Population: All Participants: Participants who consented to the study protocol. Data for participants in Cohort B with an ISWT initiated at least 1 h following completion of previous ISWT (Period 2) are presented.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Cohort B: Non-Treprostinil PAH Medications
Number analyzed (Participants) | 23
scores on a scale
  PAH, Baseline | 1.13 (0.34)
  PAH, Change at least 1 h following completion of previous ISWT (Period 2) on Day 1 | 1.87 (0.97)
  SOB, Baseline | 1.04 (0.21)
  SOB, Change at least 1 h following completion of previous ISWT (Period 2) on Day 1 | 2.13 (0.92)
  Fatigue, Baseline | 1.13 (0.34)
  Fatigue, Change at least 1 h following completion of previous ISWT (Period 2) on Day 1 | 1.91 (1.04)

5. Secondary Outcome: Change From Baseline in Modified Borg Dyspnea Scores at Day 1
Description: The modified Borg scale allows participants to rate maximum level of dyspnea experienced during 6-Minute Walk Test (6MWT). Scores ranged from 0 (best condition) to 10 (worst condition). Baseline defined as average from Borg Dyspnea Scores measured at 15 and 0 m prior to ISWT. If a single pre-ISWT Borg Dyspnea Score was missing, the other nonmissing single score was used as baseline value. Change from Baseline=Post-Baseline value - Baseline value. Data for participants in Cohort A with an ISWT initiated at 30 m of previous dose (expected peak level) and an ISWT initiated at 3-4 h of previous dose of inhaled treprostinil (expected trough level) on Day 1 are presented. Data for participants in Cohort B with an ISWT initiated at 4 h after morning dose of non-treprostinil PAH medication (Period 1) and with an ISWT initiated at least 1 h following completion of previous ISWT (Period 2) on Day 1 are presented. Peak and trough levels are highest and lowest concentrations of a drug in plasma.
Time Frame: Baseline, ~30 m of previous dose of inhaled treprostinil, ~3-4 h of previous dose of inhaled treprostinil, ~4 h after morning dose of non-treprostinil PAH medication, and ≥1 h following completion of previous ISWT on Day 1
Population: All Participants: Participants who consented to the study protocol. Here, 'Number Analyzed' signifies participants evaluable at the specified timepoint.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Cohort A: Treprostinil | Cohort B: Non-Treprostinil PAH Medications
Number analyzed (Participants) | 20 | 23
scores on a scale
  Expected peak level, Baseline: number analyzed (Participants) | 20 | 0
  Expected peak level, Baseline | 0.28 (0.54) |
  Change at 30 m of previous dose of inhaled treprostinil (expected peak level) on Day 1: number analyzed (Participants) | 20 | 0
  Change at 30 m of previous dose of inhaled treprostinil (expected peak level) on Day 1 | 3.00 (1.78) |
  Expected trough level, Baseline: number analyzed (Participants) | 20 | 0
  Expected trough level, Baseline | 0.23 (0.62) |
  Change at 3-4 h of previous dose of inhaled treprostinil (expected trough level) on Day 1: number analyzed (Participants) | 20 | 0
  Change at 3-4 h of previous dose of inhaled treprostinil (expected trough level) on Day 1 | 3.13 (2.16) |
  Period 1, Baseline: number analyzed (Participants) | 0 | 23
  Period 1, Baseline |  | 0.24 (0.50)
  Change at 4 h after morning dose of non-treprostinil PAH medication (Period 1) on Day 1: number analyzed (Participants) | 0 | 23
  Change at 4 h after morning dose of non-treprostinil PAH medication (Period 1) on Day 1 |  | 2.85 (1.81)
  Period 2, Baseline: number analyzed (Participants) | 0 | 23
  Period 2, Baseline |  | 0.23 (0.64)
  Change at least 1 h following completion of previous ISWT (Period 2) on Day 1: number analyzed (Participants) | 0 | 23
  Change at least 1 h following completion of previous ISWT (Period 2) on Day 1 |  | 3.03 (1.90)

6. Other Pre Specified Outcome: Change From Baseline in Pulse Oximetry at Day 1
Description: Pulse Oximetry includes the collection of saturation peripheral capillary oxygenation (SpO_2). Baseline was defined as the average from pulse oximetry measured at 15 minutes and 0 minute prior to the ISWT. In the case of a single, missing pre-ISWT pulse oximetry, the other non-missing single measurement would be used as baseline value. Change from Baseline = Post-Baseline value - Baseline value. Data for participants in Cohort A who had an ISWT initiated at 30 m of previous dose (expected peak level) and an ISWT initiated at 3-4 h of previous dose of inhaled treprostinil (expected trough level) on Day 1 are presented. Additionally, data for participants in Cohort B who included an ISWT initiated at 4 h after morning dose of non-treprostinil PAH medication (Period 1) and with an ISWT initiated at least 1 h following completion of previous ISWT (Period 2) on Day 1 are presented. Peak and trough levels are the highest and lowest concentrations of a drug in plasma.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent saturation (SpO_2)
Arm/Group | Cohort A: Treprostinil | Cohort B: Non-Treprostinil PAH Medications
Number analyzed (Participants) | 20 | 23
percent saturation (SpO_2)
  Expected peak level, Baseline: number analyzed (Participants) | 20 | 0
  Expected peak level, Baseline | 93.73 (2.94) |
  Change at 30 m of previous dose of inhaled treprostinil (expected peak level) on Day 1: number analyzed (Participants) | 20 | 0
  Change at 30 m of previous dose of inhaled treprostinil (expected peak level) on Day 1 | -8.13 (6.68) |
  Expected trough level, Baseline: number analyzed (Participants) | 20 | 0
  Expected trough level, Baseline | 95.15 (3.12) |
  Change at 3-4 h of previous dose of inhaled treprostinil (expected trough level) on Day 1: number analyzed (Participants) | 20 | 0
  Change at 3-4 h of previous dose of inhaled treprostinil (expected trough level) on Day 1 | -10.35 (9.35) |
  Period 1, Baseline: number analyzed (Participants) | 0 | 23
  Period 1, Baseline |  | 94.98 (3.24)
  Change at 4 h after morning dose of non-treprostinil PAH medication (Period 1) on Day 1: number analyzed (Participants) | 0 | 23
  Change at 4 h after morning dose of non-treprostinil PAH medication (Period 1) on Day 1 |  | -4.85 (5.13)
  Period 2, Baseline: number analyzed (Participants) | 0 | 23
  Period 2, Baseline |  | 94.04 (3.14)
  Change at least 1 h following completion of previous ISWT (Period 2) on Day 1: number analyzed (Participants) | 0 | 23
  Change at least 1 h following completion of previous ISWT (Period 2) on Day 1 |  | -2.91 (3.79)

7. Other Pre Specified Outcome: Change From Baseline in Heart Rate at Day 1
Description: Heart rate was captured as beats per minute (bpm). Baseline was defined as the average from pulse oximetry measured at 15 minutes and 0 minute prior to the Incremental Shuttle Walk Test (ISWT). In the case of a single, missing pre-ISWT pulse oximetry, the other non-missing single measurement would be used as baseline value. Change from Baseline = Post-Baseline value - Baseline value. Data for participants in Cohort A who had an ISWT initiated at 30 m of previous dose (expected peak level) and an ISWT initiated at 3-4 h of previous dose of inhaled treprostinil (expected trough level) on Day 1 are presented. Additionally, data for participants in Cohort B who included an ISWT initiated at 4 h after morning dose of non-treprostinil PAH medication (Period 1) and with an ISWT initiated at least 1 h following completion of previous ISWT (Period 2) on Day 1 are presented. Peak and trough levels are the highest and lowest concentrations of a drug in plasma.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Cohort A: Treprostinil | Cohort B: Non-Treprostinil PAH Medications
Number analyzed (Participants) | 20 | 23
bpm
  Expected peak level, Baseline: number analyzed (Participants) | 20 | 0
  Expected peak level, Baseline | 80.08 (11.93) |
  Change at 30 m of previous dose of inhaled treprostinil (expected peak level) on Day 1: number analyzed (Participants) | 20 | 0
  Change at 30 m of previous dose of inhaled treprostinil (expected peak level) on Day 1 | 24.48 (18.10) |
  Expected trough level, Baseline: number analyzed (Participants) | 20 | 0
  Expected trough level, Baseline | 75.58 (10.78) |
  Change at 3-4 h of previous dose of inhaled treprostinil (expected trough level) on Day 1: number analyzed (Participants) | 20 | 0
  Change at 3-4 h of previous dose of inhaled treprostinil (expected trough level) on Day 1 | 23.08 (19.10) |
  Period 1, Baseline: number analyzed (Participants) | 0 | 23
  Period 1, Baseline |  | 74.59 (11.67)
  Change at 4 h after morning dose of non-treprostinil PAH medication (Period 1) on Day 1: number analyzed (Participants) | 0 | 23
  Change at 4 h after morning dose of non-treprostinil PAH medication (Period 1) on Day 1 |  | 31.28 (13.67)
  Period 2, Baseline: number analyzed (Participants) | 0 | 23
  Period 2, Baseline |  | 75.26 (12.04)
  Change at least 1 h following completion of previous ISWT (Period 2) on Day 1: number analyzed (Participants) | 0 | 23
  Change at least 1 h following completion of previous ISWT (Period 2) on Day 1 |  | 33.39 (18.08)

ADVERSE EVENTS:
Time Frame: Baseline through Day 1 (up to at least 5 hours or at the Investigator's discretion)
Description: Safety Population: All participants who initiated an ISWT at Screening.
Arm/Group | Cohort A: Treprostinil | Cohort B: Non-Treprostinil PAH Medications
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/23
Other Adverse Events (participants affected / at risk) | 0/20 | 9/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Treprostinil (N=20) | Cohort B: Non-Treprostinil PAH Medications (N=23)
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/65/NCT03888365/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-30): https://cdn.clinicaltrials.gov/large-docs/65/NCT03888365/SAP_001.pdf